CLINICAL TRIAL: NCT03256825
Title: Rapid Urinary Tract Infection Diagnosis and Real-time Antimicrobial Stewardship Decision Support - Accuracy and Effect on Antibiotic Consumption
Brief Title: Rapid Urinary Tract Infection Diagnosis and Real-time Antimicrobial Stewardship Decision Support
Acronym: RUDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Møre og Romsdal HF (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: RUDE/01-2016
Record Dates: First submitted 2017-08-15; First posted 2017-08-22 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Urinary Tract Infections
Keywords: Diagnostic accuracy; Anti-bacterial agents; Decision support systems, clinical
MeSH Terms: conditions — Urinary Tract Infections | interventions — Rapid Diagnostic Tests

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rapid diagnostics (Other): patients admitted to medical and surgical wards with urinary tract infections at Ålesund Hospital, Moere and Romsdal, Norway. Here, rapid diagnostics alone will be implemented.
  Interventions: Diagnostic Test: Rapid diagnostics alone
- Rapid diagnostics and RADS (Other): patients admitted to medical and surgical wards with urinary tract infections at Molde Hospital, Moere and Romsdal, Norway. Here, rapid diagnostics will be implemented in conjunction with Real-time antimicrobial stewardship decision support : rapid diagnostics and RADS.
  Interventions: Diagnostic Test: Rapid diagnostics alone; Other: Real-time antimicrobial stewardship decision support

INTERVENTIONS:
Diagnostic Test: Rapid diagnostics alone — Urine samples present at the laboratory at opening on weekdays will be screened using urine flow cytometry and microscopy of centrifuged gram stained urine. Samples found positive for significant mono microbial bacteriuria will be investigated further by using direct automated phenotypic identification and antimicrobial susceptibility determination.
Other: Real-time antimicrobial stewardship decision support — A clinical microbiologist will be give RADS by phone to a designated clinician with the aim of:
  1. Switch to active treatment if non-working empirical treatment
  2. De-escalate broad spectrum empiric treatment when feasible
  3. Promote early intravenous to per oral switch
  4. Shorten treatment duration
  Other Names: RADS
  Arms: Rapid diagnostics and RADS

SUMMARY:
The study aims to assess the accuracy and impact of rapid diagnosis and rapid diagnosis decision support on different aspects of antibiotic consumption when implemented alone or together.

DETAILED DESCRIPTION:
This interventional study in two centers compares two groups with each other and with a pre-intervention control group. In group 1 rapid techniques for handling urine cultures will be the only intervention. In group 2 rapid diagnostics will be supplemented with real-time antimicrobial stewardship decision support (RADS). In each center two departments will be involved.

Urine samples present at the laboratory at opening on weekdays will be screened using urine flow cytometry and microscopy of centrifuged gram stained urine. Samples found positive for significant mono microbial bacteriuria will be investigated further by using direct automated phenotypic identification and antimicrobial susceptibility determination and screened for inclusion in the interventional study.

In one of the centers, rapid techniques will be coupled to real-time antimicrobial stewardship decision support (RADS). RADS will be given by telephone to a designated clinician with the aim of:

1. Switch to active treatment if non-working empirical treatment
2. De-escalate broad spectrum empiric treatment when feasible
3. Promote early intravenous to per oral switch
4. Shorten treatment duration

ELIGIBILITY:
Inclusion Criteria:

* Urine sample present at the laboratory weekdays
* At least 11 ml of urine in sample
* Admitted to surgical or medical ward.
* Urine sample taken on admission to hospital.
* Rapid diagnostics suggesting mono microbial growth of > 100.000 microbes/ml urine.
* Clinical and laboratory signs/symptoms of urinary tract infection at time of sample delivery.

Exclusion Criteria:

* Other simultaneous infections that warrant systemic antimicrobial therapy or surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
All-cause 30-day mortality | 30 days

SECONDARY OUTCOMES:
Adherence to guidelines for empirical therapy | Recorded at inclusion or within 30 days after admission/inclusion.
  Antibiotics given before results of microbiology diagnostics.
Total antibiotic consumption in intervention groups and control group compared | Recorded at inclusion or within 30 days after admission/inclusion.
  Total consumption of antibiotic during admission and prescribed oral antibiotics after discharge. Expressed in (DDD) "the assumed average maintenance dose per day for the drug used for its main indication in adults" / admission
Use of broad spectrum antibiotics - DDD/admission in intervention groups compared with control group. | Recorded 30 days after admission/inclusion.
Time from admission to optimal antibiotic therapy | Recorded 30 days after admission/inclusion.
  Optimal treatment is defined as the working treatment with the most narrow spectrum possible
Frequency of errors by rapid diagnostics/errors in RADS leading to non-working treatment | Recorded within 30 days after admission/inclusion.
Treatment duration - intravenous/per oral | Recorded within 30 days after admission/inclusion.
Intensive care unit length of stay | Recorded within 30 days after admission/inclusion.
Hospital length of stay | Recorded within 30 days after admission/inclusion.
Frequency of adherence to treatment suggestions given as RADS | Recorded within 30 days after admission/inclusion.
Frequency of readmission for urinary tract infection within 30 days of discharge | Recorded within 30 days after admission/inclusion.
Turnaround time of rapid diagnostic procedures compared to conventional diagnostics | Recorded within 30 days after admission/inclusion.
Accuracy of rapid diagnostic procedures compared to conventional diagnostics | Recorded within 30 days after admission/inclusion.

CONTACTS AND LOCATIONS:
Overall Officials: Einar Nilsen, MD, Principal Investigator — Møre and Romsdal Health Trust
Locations (2):
- Norway (2):
  - Ålesund Hospital, Ålesund
  - Molde Hospital, Molde

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other investigators.

REFERENCES:
- [Background] Nilsen E. Automated identification and susceptibility determination directly from blood cultures facilitates early targeted antibiotic therapy. Scand J Infect Dis. 2012 Nov;44(11):860-5. doi: 10.3109/00365548.2012.689848. Epub 2012 Jul 25. PMID 22831285